CLINICAL TRIAL: NCT01493713
Title: Phase 4 Study to Evaluate Correlation of Overall Response According to RECIST-conventional Imaging Techniques, Morphologic Response by CT, & Histopathologic Response in Patients With Hepatic Metastasis Secondary to Colorectal Cancer With Bevacizumab in Combination With XELOX
Brief Title: Correlation Between RECIST, Morphologic Response by CT- Histopathologic Response in Hepatic Metastasis Secondary to Colorectal Cancer
Acronym: AVAMET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GEMCAD-10-06
Record Dates: First submitted 2011-11-22; First posted 2011-12-16 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer; Hepatic Metastasis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab, XELOX (Experimental): Bevacizumab in combination with XELOX
  Interventions: Other: Evaluate the correlation of overall different objective response.

INTERVENTIONS:
Other: Evaluate the correlation of overall different objective response. — Evaluate the correlation of overall different objectives response. Chemotherapeutic agents: XELOX scheme (Xeloda; Oxaliplatin) Device: MDCT (MultiDetector Computed Tomography)

SUMMARY:
The purpose of this study is to to evaluate the correlation of overall objective response according to RECIST v1.1. criteria evaluated by conventional imaging techniques, morphologic response by CT, and histopathologic response in patients with resectable hepatic metastasis secondary to colorectal cancer treated with bevacizumab in combination with XELOX.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age ≥ 18 years.
3. ECOG 0-1.
4. Life expectancy of at least 12 weeks.
5. Histologic confirmation of adenocarcinoma of the colon or rectum, according to the 7th edition of the TNM classification, with evidence of liver metastases according to RECIST v 1.1 criteria (Annex V). Patients with the diagnosis of liver metastasis presenting synchronically or after a disease-free interval. The primary tumor shall have been resected previously although the inverse approach may be acceptable if the tumor is not very symptomatic. Patients in whom combined surgery of the primary tumor and metastases is planned are not eligible.
6. Availability of a tumor sample for KRAS gene determination.
7. No prior chemotherapy treatment for metastatic CRC.
8. Patients with resectable hepatic metastases of colorectal carcinoma who satisfy the following criteria:

   * ≤ 4 metastases
   * Size < 10 cm
   * Technically feasible R0 resection, with a residual liver volume of no less than 30%

   NOTE: Patients with bilateral metastases may be enrolled if they satisfy the above criteria (<4 metastases and size <10 cm).
9. Adequate bone marrow, liver and kidney function, defined as:

   * Hemoglobin ≥ 9.0 g/dl (a transfusion can be given before treatment).
   * Platelet count ≥ 100 × 109/L.
   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
   * Serum bilirubin ≤ 1.5 times higher than the upper limit of normality (ULN).
   * Alkaline phosphatase, ALT (SGPT) and AST (SGOT) ≤ 5 × ULN.
   * Serum creatinine < 1.5 x ULN or creatinine clearance ≥ 50 ml/min according to Cockcroft and Gault formula (Annex VII).
   * INR < 1.5 within the 7 days prior to the start of study treatment. aPTT < 1.5 × ULN within 7 days prior to the start of study treatment. Exception: Patients treated with complete doses of anticoagulants due to venous thromboembolism usually must have an INR value within the established range (usually 2-3). The patient must be receiving a stable dose of anticoagulant treatment before enrollment in the study.
   * Urine strip for proteinuria < 2+. If the result of the reactive strip in urine is ≥ 2+, the 24-hour urine sample must demonstrate ≤ 1 g protein in 24 hours in order to include the patient.
10. Women of childbearing potential must have a negative pregnancy test in serum or urine in the 7-day period before entering the study. Postmenopausal women must have been amenorrheic during at least 12 months. Likewise, both the men and the women who participate in this study must use effective contraceptive methods (e.g., abstinence, intrauterine device, oral contraceptives, a double barrier method or surgical sterility), beginning upon signing the informed consent form and for at least 6 months after the end of treatment or the last dose, whichever occurs first.
11. The subject must have the capacity, in the opinion of the investigator, to comply with all the procedures and examinations of study follow-up.

Exclusion Criteria:

1. Patients with non-resectable hepatic metastases at the time of enrollment.
2. Previous systemic or local treatment of metastatic disease.
3. Presence of metastatic extrahepatic disease.
4. Neo-adjuvant or adjuvant chemotherapy/radiotherapy in the 6 months prior to entering the study.
5. Use of any investigational drug in the 4 weeks before starting the study treatment.
6. Current or recent (in the 10 days prior to the first administration of the study treatment) use of acetylsalicylic acid (> 325 mg/day) or clopidogrel (75 mg/day).
7. Current presence of peripheral neuropathy = 1 (CTCAE).
8. Hypertension not properly controlled (defined as systolic pressure > 150 mm Hg and/or diastolic pressure > 100 mm Hg in repeated measurements), despite optimal medical management.
9. Previous history of hypertensive episodes or hypertensive encephalopathy.
10. CHF class II or higher of the NYHA classification.
11. History of myocardial infarction or unstable angina within the 6 months prior to starting the study treatment.
12. Significant vascular disease (e.g., aortic aneurysm requiring surgery, pulmonary embolism or recent peripheral arterial thrombosis) in the 6 months prior to the start of the study treatment.
13. History of hemoptysis (equivalent to = ½ teaspoon of red-colored blood per episode) in the month prior to the study treatment.
14. Major surgery, open surgical biopsy or significant trauma in the 4 weeks prior to the start of study treatment. Thick-needle biopsy of a major organ in the 7 days prior to entering the study. Insertion of a vascular access > 3 days before entering the study is allowed.
15. Tests or history of significant hemorrhagic diathesis or coagulation disorder (in the absence of anticoagulation).
16. History of abdominal fistula or gastrointestinal perforation in the 6 months prior to the start of study treatment.
17. Intra-abdominal acute inflammatory process.
18. Serious unhealed wounds, active ulcer or untreated bone fracture.
19. History of another neoplastic disease aside from colorectal cancer in the last 2 years prior to the start of study treatment, with the exception of basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix treated curatively.
20. Human immunodeficiency virus infection or chronic infection by the hepatitis B or C virus or presence of uncontrolled intercurrent infections, or other severe uncontrolled concomitant diseases.
21. Current grade ≥ 2 infection (CTCAE).
22. Pregnant or breast-feeding women.
23. Known allergy, suspicion of allergy, or hypersensitivity to any of the study drugs (bevacizumab, oxaliplatin, capecitabine) and/or iodide contrast agents.
24. Incapacity for oral intake.
25. Any important and uncontrolled medical, psychological, psychiatric or social problem that can interfere in the subject's participation in the study or the evaluation of the study results or represents and increased risk of complications related to the patient's treatment.
26. Patients in whom combined surgery of the primary tumor and metastases is planned are not eligible.
27. Venous Cava invasion and 2 or more hepatic venous invasion Both portal venous invasion Remanent future minor to 40% Use of portal embolization previous to hepatectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-11-16 (Actual); Primary Completion 2014-12-08 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Correlation of overall objective responses evaluated by conventional imaging techniques with the morphologic response evaluated by MDCT and the histopathologic response after the resection of hepatic metastases. | 2016

SECONDARY OUTCOMES:
R0/R1/R2 resectability rate. | 2016
Progression-free survival (PFS), only in patients who do not undergo metastasis resection. | 2016
Recurrence-free survival (RFS) in patients who undergo metastasis resection. | 2016
Safety and toxicity (surgical and therapeutic) of the therapy graded according to CTC v.4.0 | 2016
Overall survival (OS) at 2 and 3 years. | 2016
Examine the influence of a potential predictive and prognostic tumour biomarker -mutations in K-RAS- after start of therapy on overall objective response | 2016
Examine the influence of a potential predictive and prognostic tumour biomarker -mutations in K-RAS- after start of therapy on surgical resection rate | 2016
Examine the influence of a potential predictive and prognostic tumour biomarker -mutations in K-RAS- after start of therapy on survival | 2016
Examine the influence of a potential predictive and prognostic tumour biomarker -mutations in K-RAS- after start of therapy on progression free survival | 2016

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Vera, Dr, Study Director — Hospital de Navarra
Locations (21):
- Spain (21):
  - Hospital de Donostia, San Sebastián, Guipúzcoa
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital Son Llatzer, Palma de Mallorca, Mallorca
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clìnic, Barcelona
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Complejo Hospitalario Xeral Calde, Lugo
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital de Sabadell, Sabadell
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No